# Exploring Enrollment and Participation Patterns in Weight Loss Clinical Trials Patients: An Observational Clinical Trial Perspective

This is an Informed Consent Form For Weight Loss Patients in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: November 24, 2023

### About the Informed Consent Form

The invitation to accomplish this form indicates your eligibility for prospective participation in a novel observational clinical study aimed at those suffering from weight loss. This thorough paper outlines the study's key objectives, the applied research technique, and the prospective consequences, which include both positive and potentially negative effects. Before making a choice, it's critical to fully understand the possible consequences of your engagement, and consulting with your healthcare physician can help. If any aspect of this material is unclear or if you have any queries, please contact the researcher or the appropriate people.

# Exploring the Role of Clinical Trials in Addressing Weight Loss

Weight loss refers to the reduction of body weight, typically resulting from a conscious effort to improve fitness or health. It can occur intentionally through changes in diet, increased physical activity, or lifestyle modifications, or it can be unintentional due to an underlying health condition.

Clinical trials focusing on weight loss hold substantial value in assessing the safety and effectiveness of emerging therapies for this condition. These trials act as crucial

benchmarks in determining whether new medications excel beyond established treatments, offering robust evidence to advocate for their broader utilization.

This study stands apart by placing significant focus on delving into the personal experiences of individuals grappling with weight loss, actively participating in a clinical trial involving medical interventions. The principal aim lies in meticulously analyzing both trial completion rates and instances of voluntary withdrawal within this specific group of patients.

## Emphasizing the Value of Observational Clinical Trials

Engaging in this medical trial encompasses participation in an observational study, an indispensable component of clinical research designed to glean insights through unobtrusive monitoring of patients as they adhere to their treatment routines.

Researchers will solely observe your experiences, meticulously evaluating the consequences of your condition while maintaining the integrity of your treatment regimen. This trial framework is instrumental in enhancing our understanding of the natural evolution of a specific medical condition and its implications for individuals affected by it. Your voluntary participation in this observational study plays a pivotal role in advancing medical knowledge and refining care for individuals facing similar health circumstances.

# Differentiating This Study from Other Weight Loss Clinical Trials

Recognizing the unique framework of this research study is pivotal. It operates solely on an observational basis, indicating that your engagement won't involve specific therapies or interventions. To make an informed decision about potential participation in a clinical trial, understanding the scope of weight loss clinical research, including interventional studies involving diverse treatment regimens, is crucial.

Crafting an informed decision about your potential participation in a clinical trial demands an active approach involving thorough research and comparison among trials. Platforms such as ClinicalTrials.gov provide extensive information about <u>weight loss</u> <u>studies</u>. Additionally, Power's specialized online hub offers a comprehensive compilation of ongoing <u>weight loss clinical trials</u> actively seeking participants. Through diligent exploration and a comprehensive understanding of diverse clinical trial formats, you can confidently determine your potential involvement.

### Ensuring Data Anonymity Throughout the Study

Ensuring the complete confidentiality of your information is pivotal in this study. To maintain your anonymity, kindly avoid disclosing any personal or identifiable details in your responses to the questionnaires. The devoted research team is resolute in their efforts to fortify the security and privacy of your data. However, it's crucial to acknowledge that specific legal circumstances may require the revelation of personal information.

### Actively Contributing to Clinical Trial Surveys

We want you to participate actively in this observational clinical study by contributing your views and experiences. Your involvement entails completing surveys every two weeks, which usually take 20-30 minutes. Furthermore, our staff is committed to performing quarterly check-in calls to assure continual support and your continued participation during the trial.

It is critical to emphasize that your participation in this trial's survey phase is totally optional. You have the option of answering selected questions or completing the full questionnaire based on your preferences. Moreover, you retain the right to withdraw from the trial at any stage. Recognizing the personal significance of participating in a clinical research, we pledge to provide the necessary assistance, protect your privacy, and guide your choice.

# Health Implications and Risks

While clinical trials have brought about significant advancements, comprehending potential health repercussions for participants, notably in studies involving drug evaluation, remains pivotal.

Nonetheless, in observational clinical research, we adopt a distinct approach to minimize these impacts by abstaining from providing experimental drugs to participants. Our core focus is on meticulous monitoring and evaluating outcomes to ensure the prevention of any avoidable health risks.

### **Expected Benefits**

While participants in this observational clinical research might not experience immediate benefits, their involvement could bear significant long-term implications. The data gathered from participants will aid in developing future approaches for engaging individuals dealing with weight loss, potentially broadening avenues for medical research. Those participating in this clinical trial have the potential to drive substantial progress in the field of medical research, potentially paving the way for future weight loss patients.

### More to Read on Diversity in Clinical Studies

To explore the intricate landscape of diversity within clinical trials, numerous online resources are available to deepen your comprehension.

Whether you aim to grasp the complexities of challenges and possibilities related to diversity in clinical trials or broaden your personal perspectives, these resources can serve as valuable tools:

Reopell, Luiza, Timiya S. Nolan, Darrell M. Gray, Amaris Williams, LaPrincess C. Brewer, Ashley Leak Bryant, Gerren Wilson et al. "Community engagement and clinical trial diversity: Navigating barriers and co-designing solutions—A report from the "Health Equity through Diversity" seminar series." *PloS one* 18, no. 2 (2023): e0281940.

Marrie, Ruth Ann, Jeremy Chataway, Barbara E. Bierer, Marcia Finlayson, Elena H. Martinez-Lapiscina, Jennifer Panagoulias, Maria Pia Sormani, Mitzi Joi Williams, and Lilyana Amezcua. "Enhancing diversity of clinical trial populations in multiple sclerosis." *Multiple Sclerosis Journal* 29, no. 9 (2023): 1174-1185.

# Confirmation of Participant

I verify that I've dedicated sufficient time to comprehend and absorb the information within the informed consent form, either through self-review or with the guidance of

| professionals who explained its contents. I adequately resolved. | 'm content that all my inquiries have been |
|---|---|
| Participant Name | |
| Participant Signature | |
| Date | |
| Confirmation of Facilitator | |
| I assert that I engaged in a thorough converse elaborating on the intricacies detailed in the participant's complete grasp of the princutilized, potential risks and benefits, and or clinical trial. | is written document. My aim was to ensure nary research objectives, methodology |
| Printed Name of Assisting Researcher | |
| Signature of Assisting Researcher | |
| Date | |